CLINICAL TRIAL: NCT07098650
Title: Haemdall: Developing a Quantitative MRI Biomarker of Classical (Infratentorial) Superficial Siderosis of the Central Nervous System
Brief Title: Haemdall: Developing a Quantitative MRI Biomarker of Infratentorial Superficial Siderosis of the Central Nervous System
Acronym: Haemdall
Status: Recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: 24/PR/1441
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Superficial Siderosis
Keywords: brain iron; MRI; Quantitative Susceptibility Mapping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Superficial siderosis cohort: Individuals diagnosed with infratentorial superficial siderosis
- Healthy volunteer cohort: Healthy volunteers without other neurological condition or significant disease

SUMMARY:
Haemdall: Using Medical Imaging to measure Brain Iron in Superficial Siderosis.

This study is looking at a new way of using MRI scans to potentially measure the amount of iron on the surface of the brain. Iron build up in the brain is linked to how superficial siderosis develops. The study will also aim to see if there is a connection between the amount of iron in the brain and common superficial siderosis symptoms. Clinical tests will be used to measure symptoms including tests to measure your hearing, walking & balance and participants' ability to remember, think and understand.

ELIGIBILITY:
Inclusion Criteria:

Superficial siderosis cohort:

* Male or female adults of 18 years of age or older with a confirmed diagnosis of superficial siderosis
* Participants who have the capacity and a level of English proficiency that allows him/her to communicate well with the Investigator, understand and comply with the requirements of the investigation, read all participant facing documentation, as well as read and sign the informed consent form.
* Participants willing and able to give informed consent for participation in the investigation

Healthy cohort:

* Male or female over 18 years of age without a diagnosis of a neurological disorder
* Participants who have the capacity and a level of English proficiency that allows him/her to communicate well with the Investigator, understand and comply with the requirements of the investigation, read all participant facing documentation, as well as read and sign the informed consent form.
* Participants willing and able to give informed consent for participation in the investigation

Exclusion Criteria:

* The participant may not enter the investigation if they have any contraindication to magnetic resonance imaging (including pregnancy, extensive tattoos, pacemaker, shrapnel injury or metallic unfixed implanted devices, metallic fragments, severe claustrophobia and cochlear implants)
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the investigation, or may influence the result of the investigation, or the participant's ability to participate in the investigation
* Participants who do not demonstrate the capacity to understand the investigation information or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 participants from around the UK
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association and clinical relevance of with markers of neurodegeneration and clinical assessments | through study completion, an average of 1 year
  1. Correlation between magnetic susceptibility assessed by QSM and brain cognitive function by MoCA.
  2. Correlations between magnetic susceptibility assessed by QSM and: a) markers of neurodegeneration; and b) clinical assessment outcomes (auditory, balance, gait, cognitive)

SECONDARY OUTCOMES:
Radiologist observational scoring and test-retest | through study completion, an average of 1 year
  1. The agreement between radiologist scored observational level of iron accumulation via the Queens Square Superficial Siderosis (QUASARS) rating scale and quantitative MRI measure related to iron on the brain surface. The QUASARS rating is out of 36 points; with higher scores indicate a worse outcome
  2. The repeatability coefficient within a single scanning session

CONTACTS AND LOCATIONS:
Locations (1):
- Perspectum, Oxford, United Kingdom